CLINICAL TRIAL: NCT05822882
Title: Efficacy of Postoperative Epidural Anesthesia Following Abdominoplasty
Acronym: EDA
Status: Completed | Type: Observational
Sponsor: Klinik Bogenhausen (Other)
Collaborators: ISAR Klinikum (Other)
Responsible Party: Principal Investigator, Ulf Dornseifer, MD, Principal Investigator, ISAR Klinikum
Other Study IDs: EDA following Abdominoplasty
Record Dates: First submitted 2023-03-11; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Abdominoplasty
Keywords: abdominoplasty; postoperative analgesia; regional anesthesia; epidural anesthesia; epidural catheter
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with epidural anesthesia: Patients following Abdominoplasty with postoperative epidural anesthesia via pain catheter
  Interventions: Procedure: Epidural anesthesia
- Patients without epidural anesthesia: Patients following Abdominoplasty without postoperative epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — Postoperative pain management by epidural anesthesia via epidural catheter and pain pump
  Groups: Patients with epidural anesthesia

SUMMARY:
Effective postoperative pain management is essential for patient satisfaction and therefore intraoperative regional nerve blocks have become more and more popular in abdominoplasties. However, the key disadvantage of these blocks are their limited duration of action. This observational study evaluates the effects of a longer- lasting, individualized epidural analgesia using a pain pump to better classify the clinical value of this procedure.

DETAILED DESCRIPTION:
This work reviews the digital medical charts of patients who underwent selective abdominoplasty without additive surgical procedures within a period of 4 years. Evaluated data comprise the postoperative analgesia regimen, including on-demand medication, mobilization time, inpatient length of stay, and clinical outcome. The patients were grouped by the presence of an epidural catheter.

ELIGIBILITY:
Inclusion Criteria:

• Patients who underwent abdominoplasty

Exclusion Criteria:

• Patients who underwent abdominoplasty combined with additional intraoperative procedures (e.g., liposuction, hernia repair) were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent abdominoplasty at the Department of Plastic Surgery, ISAR Klinikum, Munich, Germany, between September 2018 and August 2022
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
frequency of retrieval of the on-demand non-epidural opiate | from the day of inpatient admission to the day of discharge of every included patient. The event determined by reviewing digital medical charts, is therefore assessed for an estimated period of up to 7 days
  frequency of retrieval of the on-demand non-epidural opiate as a measure of perceived pain discomfort

SECONDARY OUTCOMES:
postoperative mobilization ability | from the day of inpatient admission to the day of discharge of every included patient. The event determined by reviewing digital medical charts, is therefore assessed for an estimated period of up to 7 days
  the time at which the patient was able to move at room level with the assistance of a nurse (assisted full mobilization), the time at which the patient was able to get out of bed independently and move without assistance (independent full mobilization)
timing of urinary catheter removal | from the day of inpatient admission to the day of discharge of every included patient. The event determined by reviewing digital medical charts, is therefore assessed for an estimated period of up to 7 days
  timing of urinary catheter removal after surgery
length of hospital stay | from the day of inpatient admission to the day of discharge of every included patient. The event determined by reviewing digital medical charts, is therefore assessed for an estimated period of up to 7 days
  number of days from the day of surgery until dischargement

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Dornseifer, MD, Principal Investigator — ISAR Klinikum
Locations (1):
- ISAR Klinikum, München, Bavaria, Germany